CLINICAL TRIAL: NCT00599560
Title: Vasopressin and V2 Receptor in Meniere's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osaka University (Other)
Collaborators: Osaka City University (Other)
Responsible Party: Meniere's disease association at Osaka University, Tadashi Kitahara, M.D.,Ph.D.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: tk19661218; Osaka Univ. School of Medicine
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2008-01

CONDITIONS: Meniere Disease
Keywords: Meniere's disease; stress; vasopressin; endolymphatic sac; V2 receptor; cyclic AMP; Plasma vasopressin level and V2R mRNA expression level in the endolymphatic sac both were significantly higher in patients with Meniere's disease.; In Meniere's disease, there were significant negative co-relationships between vasopressin and V2R.; The cyclic AMP activity was basically up-regulated in the endolymphatic sac in Meniere's disease..; The cyclic AMP sensitivity for vasopressin was significantly elevated in the endolymphatic sac in Meniere's disease.
MeSH Terms: conditions — Meniere Disease; Diabetes Insipidus; Diabetes Insipidus, Nephrogenic | interventions — Vasopressins; Receptors, Vasopressin; Cyclic AMP

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Meniere's disease (Experimental): Patients were eligible for enrollment if they had received a clinical diagnosis of Meniere's disease according to the 1995 AAO-HNS criteria (Committee, 1995). These criteria can be briefly described as follows: 1) Repeated attacks of vertigo: A definitive spell is spontaneous vertigo lasting at least 20 minutes. A mixed type of spontaneous nystagmus is observed during attacks. 2) Fluctuating cochlear symptoms: The hearing test usually reveals a marked fluctuation of the threshold in the low and middle tone range.
  Interventions: Genetic: vasopressin, V2 receptor and cyclic AMP
- 2. Acoustic neurinoma (No Intervention): Diagnosed by CT and/or MRI

INTERVENTIONS:
Genetic: vasopressin, V2 receptor and cyclic AMP — plasma vasopressin, V2 receptor, cyclic AMP
  Other Names: plasma vasopressin; V2 receptor; cyclic AMP
  Arms: 1. Meniere's disease

SUMMARY:
Summary: Some of sicknesses are well known to be provoked by inadequate adaptation to physical and/or psychogenic stress in their daily life. Meniere's disease is also a common inner ear disease accompanied with vertigo, hearing loss and tinnitus especially in civilized people under stressed life style. Its oto-pathology was firstly revealed in 1938 to be inner ear endolymphatic hydrops through the temporal bone study. To elucidate the neuroscientific relationship between "stress" and "inner ear", we examined plasma vasopressin (the anti-diuretic "stress" hormone) and its receptor, V2R in the endolymphatic sac (the "inner ear" endo-organ for endolymph absorption) in Meniere's patients.

DETAILED DESCRIPTION:
Methods: Between 1998 and 2006, we enrolled and assigned 105 intractable Meniere's patients to examine plasma vasopressin during remission of vertigo attacks (controls: 30 patients with chronic otitis media). Using the real-time PCR method, we examined V2R mRNA expression in the endolymphatic sac in 12 patients (controls: 6 patients with acoustic neurinoma). By means of cell culture and cyclic AMP assay, we also examined cyclic AMP activity in the endolymphatic sac in 3 patients (controls: 3 patients with acoustic neurinoma).

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for enrollment if they had received a clinical diagnosis of Meniere's disease according to the 1995 AAO-HNS criteria (Committee, 1995). These criteria can be briefly described as follows:

  1. Repeated attacks of vertigo: A definitive spell is spontaneous vertigo lasting at least 20 minutes. A mixed type of spontaneous nystagmus is observed during attacks.
  2. Fluctuating cochlear symptoms: The hearing test usually reveals a marked fluctuation of the threshold in the low and middle tone range.

Exclusion Criteria:

* Any other neuro-otologic diseases.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 1998-04; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
plasma vasopressin level and V2 receptor mRNA in the endolymphatic sac in Meniere's disease vs controls | prospective

SECONDARY OUTCOMES:
cyclic AMP activity in the endolymphatic sac in Meniere's disease vs controls | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Kitahara, M.D.,Ph.D., Principal Investigator — Department of ORL, Osaka University, School of Medicine; Hiroshi Kiyama, Ph.D., Study Director — Department of Neuroanatomy, Osaka City University, School of Medicine; Takeshi Kubo, M.D.,Ph.D., Study Chair — Department of ORL, Osaka University, School of Medicine
Locations (1):
- Department of Otolaryngology, Osaka University, School of Medicine, Suita, Osaka, Japan

REFERENCES:
- [Result] Kumagami H, Beitz E, Wild K, Zenner HP, Ruppersberg JP, Schultz JE. Expression pattern of adenylyl cyclase isoforms in the inner ear of the rat by RT-PCR and immunochemical localization of calcineurin in the organ of Corti. Hear Res. 1999 Jun;132(1-2):69-75. doi: 10.1016/s0378-5955(99)00035-0. PMID 10392549
- See also: Meniere's disease group at Department of ORL, Osaka University, School of Medicine — http://www.med.osaka-u.ac.jp/pub/ent/r_vertigo.html